CLINICAL TRIAL: NCT00153959
Title: Psychiatric Day Hospital Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: QLG4-CT-2000-01700
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Depressive Disorders; Schizophrenia; Anxiety Disorders; Personality Disorders; Adjustment Disorders
MeSH Terms: conditions — Depressive Disorder; Schizophrenia; Anxiety Disorders; Personality Disorders; Adjustment Disorders

INTERVENTIONS:
Behavioral: acute psychiatric day care

SUMMARY:
The aim of the study was to compare the effectiveness of acute psychiatric day care to conventional inpatient care within a cross-national multi-site randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have presented with a mental disorder with current symptoms that had either led to at least a moderate disturbance in performance in more than one area of daily living or had jeopardized the residential, financial or occupational status of the patient or his family
* Treatments other than inpatient or day hospital care must have been inadequate or not sufficiently effective for the patient's current mental state

Exclusion Criteria:

* Temporary admission for diagnostic purposes or for other reasons
* Under 18 or over 65 years
* Admission without consent of the patient (according to country-specific legal regulations)
* One-way journey to hospital longer than 60 minutes
* Suicidal risk
* Risk to others
* Degree of severity of the disorder requires measures restrictive of the patient's freedom on the day of admission, or a 1:1 supervision, or deems such probable
* Acute intoxication
* Main clinical diagnosis: addictive disorder
* Presence of a somatic disorder requiring inpatient care
* Direct transfer from a different hospital
* Homelessness
* Need for constant pick-up and delivery service
* Inability to give informed consent with respect to participating in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W. Kallert, Prof.Dr., Principal Investigator — Department of Psychiatry at Dresden University of Technology
Locations (5):
- Department of Psychiatry, First Medical Faculty, Charles University of Prague, Prague, Czechia
- Department of Psychiatry at Dresden University of Technology, Dresden, Saxony, Germany
- Department of Psychiatry, Wroclaw University of Medicine, Wroclaw, Poland
- Michalovce Psychiatric Hospital, Michalovce, Slovakia
- Unit for Social and Community Psychiatry, Barts' and The London School of Medicine, London, United Kingdom

REFERENCES:
- [Derived] Gibbon S, Khalifa NR, Cheung NH, Vollm BA, McCarthy L. Psychological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007668. doi: 10.1002/14651858.CD007668.pub3. PMID 32880104
- [Derived] Kallert TW, Priebe S, McCabe R, Kiejna A, Rymaszewska J, Nawka P, Ocvar L, Raboch J, Starkova-Kalisova L, Koch R, Schutzwohl M. Are day hospitals effective for acutely ill psychiatric patients? A European multicenter randomized controlled trial. J Clin Psychiatry. 2007 Feb;68(2):278-87. doi: 10.4088/jcp.v68n0214. PMID 17335327